CLINICAL TRIAL: NCT06133179
Title: Pilot Study of the Characterization of Subacute Ischemic Cerebrovascular Accidents in the Region of the Middle Cerebral Artery by 3D Ultrasound Localization Microscopy (ULM) with a Research Ultrasound System and Non-marketed 2D Matrix Probe.
Brief Title: Super-Resolution Ultrasound of the Brain in 3D
Acronym: ESRC3D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP230511
Record Dates: First submitted 2023-10-27; First posted 2023-11-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Stroke
MeSH Terms: conditions — Stroke | interventions — contrast agent BR1

STUDY DESIGN:
Intervention Model Description: Proof of concept, exploratory, single group, non-comparative, uncontrolled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort group (Experimental): Routine care + transtemporal ultrasound examination with contract product during hospitalization
  Interventions: Procedure: Transtemporal ultrasound with contrast product (Sonovue)

INTERVENTIONS:
Procedure: Transtemporal ultrasound with contrast product (Sonovue) — During their hospitalization and in the 7 days following their stroke, all patients will perform a transtemporal ultrasound including the use of Sonovue contrast product.
  The examination will last 1 hour and will be carried out on the opposite side of the stroke then on the side of the stroke

SUMMARY:
The goal of this proof of concept study is to determine if the visualization of the middle cerebral artery and its perforators, through 3D transtemporal ultrasound imaging, is possible thanks to an off-line analysis by 3D ultrasound localization microscopy. Visualization of these vessels would allow us to conclude on the presence, or absence, of an ischemic stroke in the region of the middle cerebral artery.

To answer the question asked, 20 participants who suffered a stroke will carry out a transtemporal ultrasound examination specifically for research in the 7 days following his stroke. The data obtained will be analyzed by the CNRS medical imaging laboratory, in order to characterize the presence of a stroke and to compare the data obtained with that of standard examinations (CT and MRI).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over
* Hospitalized patient with ischemic stroke in the deep territory of the middle cerebral artery
* Patient with lesion observable on MRI
* Patient included between 24 hours and 7 days after the ischemic stroke
* Patient with a temporal window which allows soundproofing of the polygon of Willis and the middle cerebral artery
* Patient having signed free, informed and written consent
* Patient affiliated to a social security system (excluding AME)

Exclusion Criteria:

* Contralateral middle cerebral artery territory stroke or contralateral middle cerebral artery occlusion
* Patient with contraindication to Doppler ultrasound with contrast (right-left shunt, severe pulmonary arterial hypertension)
* Patient with hypersensitivity to the active princip of Sonovue (sulfur hexafluoride) or these excipients
* Patient with uncontrolled systemic hypertension
* Patient with respiratory distress syndrome
* Patient under guardianship or curatorship
* Pregnant or breastfeeding patient (positive blood pregnancy test during hospitalization)
* Patient with damaged skin at the temporal level
* Patient having presented in the 7 days preceding inclusion an acute coronary syndrome or suffering from unstable ischemic heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Describe the vascular mapping obtained by 3D transcranial ULM of patients with ischemic stroke in the territory of the middle cerebral artery and its perforators | Day 1
  Measure of the caliber of visible vessels (mm)
Describe the vascular mapping obtained by 3D transcranial ULM of patients with ischemic stroke in the territory of the middle cerebral artery and its perforators | Day 1
  Measure of the number of visible vessels (number)
Describe the vascular mapping obtained by 3D transcranial ULM of patients with ischemic stroke in the territory of the middle cerebral artery and its perforators | Day 1
  Measure of the speed of the flows (mm/sec)
Describe the vascular mapping obtained by 3D transcranial ULM of patients with ischemic stroke in the territory of the middle cerebral artery and its perforators | Day 1
  Measure of the directionality of the flows
Describe the vascular mapping obtained by 3D transcranial ULM of patients with ischemic stroke in the territory of the middle cerebral artery and its perforators | Day 1
  Measure of the diffusion index

SECONDARY OUTCOMES:
Compare 3D ULM with standard stroke imaging methods (TOF MRI and DWI) | Day 1
  vessels caliber (mm)
Compare 3D ULM with standard stroke imaging methods (TOF MRI and DWI) | Day 1
  visible vessels (number)
Compare 3D ULM with standard stroke imaging methods (TOF MRI and DWI) | Day 1
  stroke size (mm3)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Bichat, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No